CLINICAL TRIAL: NCT02684682
Title: Effect of Self-performed Mechanical Control of Plaque Frequency in Patients With Historic of Periodontitis and in Maintenance
Brief Title: Frequency of Self-performed Mechanical Control of Plaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Juliana Maier, Master in dental science with an emphasis on periodontics, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 50208115.9.0000.5346
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Gingivitis; Oral Health
Keywords: Toothbrushing; Gingivitis; Dental Plaque; Periodontal Diseases; Clinical Trial
MeSH Terms: conditions — Gingivitis; Dental Plaque; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 12h Group (Other): Intervention 'Frequency of mechanical control of plaque (12h)'
  Interventions: Behavioral: Frequency of mechanical control of plaque (12h)
- 24h Group (Other): Intervention 'Frequency of mechanical control of plaque (24h)'
  Interventions: Behavioral: Frequency of mechanical control of plaque (24h)
- 48h Group (Other): Intervention 'Frequency of mechanical control of plaque (48h)'
  Interventions: Behavioral: Frequency of mechanical control of plaque (48h)

INTERVENTIONS:
Behavioral: Frequency of mechanical control of plaque (12h) — Performing oral hygiene 12 in 12 hours, with tooth brush and interdental device.
  Arms: 12h Group
Behavioral: Frequency of mechanical control of plaque (24h) — Performing oral hygiene 24 in 24 hours, , with tooth brush and interdental device.
  Arms: 24h Group
Behavioral: Frequency of mechanical control of plaque (48h) — Performing oral hygiene 48 in 48 hours, , with tooth brush and interdental device.
  Arms: 48h Group

SUMMARY:
The purpose of this blind randomized clinical trial is to evaluate different frequencies in self-mechanical control of plaque in individuals with historic of periodontitis and in periodic and preventive maintenance in order to assess which frequencies are compatible with maintaining gingival health.

DETAILED DESCRIPTION:
Thirty nine subjects with at most 5% of the sites for GI= 2 (gingival health) will be randomized into three groups with different frequencies in self-mechanical control of plaque: Group 12 hours, 24 hours and 48 hours. The exams of plaque index, gingival index, probing depth, bleeding on probing, clinical attachment level and gingival crevicular fluid will be performed at baseline, 15, 30, 60 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with historic of periodontitis (loss of interproximal insertion ≥3mm in two or more non-adjacent teeth) treated in the Clinic of Postgraduate Periodontics at the Federal University of Santa Maria and included in the periodontal maintenance program;
* Minimum age of 35;
* Individuals with at least 12 teeth in the mouth;
* Maximum of 15% of sites with gingivitis;
* Maximum of 25% of sites with bleeding on probing.

Exclusion Criteria:

* Smokers;
* Pregnant women;
* Individuals with dryness of the mouth (xerostomia);
* Diabetics;
* Psychomotor disturbances;
* Orthodontic equipment;
* Antimicrobial prophylaxis;
* Individuals using any medication associated with gingival overgrowth;
* Individuals that used antibiotic/anti -inflammatory in recent 3 months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline gingival index at 30, 60 and 90 days. | 30,60 and 90 days.
  Assess how different frequencies of self-performed mechanical control of plaque interfere in gingival status.

SECONDARY OUTCOMES:
Changes from baseline plaque level at 30,60 and 90 days. | 30,60 and 90 days.
  * Assess how different frequencies of self-performed mechanical control of plaque interfere in the accumulation of supragingival biofilm.
  * Correlate changes in plaque levels with changes in gingival index.
Changes from volume of gingival fluid at 30,60 and 90 days. | 30,60 and 90 days.
  * Assess how different frequencies of self-performed mechanical control of plaque interfere in the volume of gingival fluid.
  * Correlate volume of gingival fluid with GI scores and bleeding on probing scores.

CONTACTS AND LOCATIONS:
Overall Officials: Karla Z Kantorski, Study Director — Universidade Federal de Santa Maria
Locations (1):
- Juliana Maier, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reiniger APP, Maier J, Wikesjo UME, Moreira CHC, Kantorski KZ. Correlation between dental plaque accumulation and gingival health in periodontal maintenance patients using short or extended personal oral hygiene intervals. J Clin Periodontol. 2021 Jun;48(6):834-842. doi: 10.1111/jcpe.13448. Epub 2021 Mar 23. PMID 33751652
- [Derived] Maier J, Reiniger APP, Sfreddo CS, Wikesjo UM, Kantorski KZ, Moreira CHC. Effect of self-performed mechanical plaque control frequency on gingival health in subjects with a history of periodontitis: A Randomized Clinical Trial. J Clin Periodontol. 2020 Jul;47(7):834-841. doi: 10.1111/jcpe.13297. Epub 2020 May 20. PMID 32315448